CLINICAL TRIAL: NCT04698720
Title: Contribution of Psychological Factors in the Healing of the Diabetic Foot Ulcer, in Physiological Indicators of Healing Prognosis and Quality of Life: a Randomized Longitudinal Trial With a Nested Qualitative Study of Effectiveness Assessment
Brief Title: Contribution of Psychological Factors in the Healing of the Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Maria da Graça Pereira, Associate Professor with Aggregation of School of Psychology, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTCD/PSIGER/ 28163/2017
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Ulcer Healing; Quality of Life; Hypnosis; Relaxation
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Muscle Relaxation; Imagery, Psychotherapy; Hypnosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment This is a Randomized Controlled Study of a Psychological Intervention (Grant et al., 2018). This study will use a mixed-methods approach nested in a 4-arm randomized control design. Qualitative and quantitative data will be collected in order to provide better understanding about the effectiveness of the hypnosis intervention in patients with DFU.
  Participants will be randomised at a ratio of 1:1 for the four conditions - EG1, EG2, ACG and PCG; and will be evaluated on the day of the first chronic DFU appointment or nursing treatment (T0), two months later (at the end of the intervention in EG, EG2, and ACG; T1), as well as six months later (T2) in a follow-up evaluation. Participants from all four groups will undergo standard treatment for the DFU, according to the guidelines of the Portuguese General Health Direction (DGS, 2010) and the International Working Group on the Diabetic Foot (IWGDF, 2015).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) Eligible participants will be randomized into the four groups into blocks of variable size, multiples of three; and will be stratified according to: i) data collection site; ii) Chronic Renal Disease (CRD); and iii) Peripheral Arterial Disease (PAD); since CRD and PAD are factors of poor prognosis in the DFU healing (Ferreira et al., 2014). This procedure will be performed using an online random number generator by an independent researcher unaware of the numeric coding for each group. After this procedure, it will not be possible to conceal the group to which the patient belongs from the researcher that will perform the psychological and placebo interventions. However, health professionals will be blinded during the entire procedure as they will only fill in the clinical questionnaire (doctors) and the RESVECH 2.0 (nurses), which assesses the DFU healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Muscle Relaxation with Guided Imagery (Experimental): Participants in the Experimental Group 1 will receive four individual 45-minute sessions, every two weeks, of progressive muscle relaxation intervention with guided imagery focused on ulcer healing, carried out by the Psychologist responsible for implementing the project, on the day of the Diabetic Foot appointments.
  Interventions: Behavioral: Muscle Relaxation with Guided Imagery
- Hypnosis with Guided imagery (Experimental): Participants in the Experimental Group 2 will receive a four individual 45-minute sessions, every two weeks, of hypnosis intervention with guided imagery focused on ulcer healing, carried out by the qualified Hypnotherapists external to the research study, on the day of the Diabetic Foot appointments.
  Interventions: Behavioral: Hypnosis with Guided Imagery
- Active Control Group (Placebo Comparator): Participants in the ACG will receive four individual 45-minute sessions of neutral guided imagery placebo focused on the patient's life before the foot ulcer, carried out by the Psychologist responsible for implementing the project, on the day of the Diabetic Foot appointments.
  Interventions: Behavioral: Neutral Guided Imagery
- Passive Control Group (No Intervention): Participants in the PCG will not receive any intervention or placebo session.

INTERVENTIONS:
Behavioral: Muscle Relaxation with Guided Imagery — Relaxation intervention session begins with diaphragmatic breathing, followed by Jacobson's progressive muscle relaxation, which involves the contraction and subsequent relaxation of the 16 muscle groups of the body (forearm, arm, upper forehead, eye, mouth, jaw and throat, neck, shoulder, chest, stomach, thigh, leg and foot).The contraction is performed for 7 seconds while the relaxation lasts for about 40 to 50 seconds.The relaxation of the foot muscle group is only performed on the healthy foot, because dressing and bandages may bandage the foot with the DFU, which together with the typical joint stiffness of the diabetic foot, make it difficult to perform. After muscle relaxation, begins the guided imagery focused on DFU healing. The patient is instructed to think about his/her current state of health and to imagine the DFU as a dark area and the healing relaxation as a light associated to pleasant sensations, which will focus on the foot with DFU to heal it.
  Arms: Muscle Relaxation with Guided Imagery
Behavioral: Hypnosis with Guided Imagery — In the beginning of the first session we apply the Eye-Roll Test for Hypnotizability of Herbert Spiegel. Each session follows the Hypnotic Protocol with the following steps:Pre-talk/Absortion/Ratification/Aliciation/Dissociation/Awakening.
  The four sessions train the participants in visual, auditory and kinesthetic perception on ulcer healing. The protocol also promotes medical treatment acceptance.
  Arms: Hypnosis with Guided imagery
Behavioral: Neutral Guided Imagery — This placebo consists of neutral guided imagery focused on themes of the patient's daily life before having DFU. Each session has a theme associated with the patient's life - family, work, friends, and leisure. Initially, the patient is asked to think about an event related to the theme of the session of his/her choice, positive or negative, which occurred before patient has the current DFU. Then, the patient is asked about a number of questions regarding the chosen episode in order to promote a more detailed reconstruction of the event. The patient is asked to imagine according to the instructions given by the Psychologist. When the whole episode is remembered, the patient is asked to tell what he or she imagined/remembered regarding each of the questions.
  Arms: Active Control Group

SUMMARY:
Diabetic foot ulcers (DFU) are one of the most serious complications of diabetes and can lead to amputations in 85% of cases, resulting in physical, psychological, family, social and economic consequences. Research suggests that psychological factors may play an important role in DFU healing. Relaxation and hypnosis seem to contribute to faster wound healing. More research is needed to assess the effectiveness of different types of intervention on different types of wounds, in particular chronic wounds such as DFU.

This study will evaluate the efficacy of relaxation and hypnosis, both with guided imagery, in DFU healing, physiological indicators (inflammatory, metabolic, oxidative stress, angiogenic, and miRNA biomarkers) of wound healing prognosis, and QoL, in patients with diabetic foot and a chronic ulcer. This study is a Randomized Controlled Study of a Psychological Intervention that aims to evaluate the efficiency of a muscle relaxation intervention with guided imagery (experimental group - EG1) compare to a hypnosis intervention with guided imagery (experimental group - EG2) and a neutral guided imagery placebo (active control group - ACG) and a group that does not receive any psychological intervention (passive control group - PCG).

This study will also examine, qualitatively, the perspectives of patients with DFU on the relaxation and hypnosis interventions, in order to check its effectiveness; as well as the perspectives of informal caregivers on this adjuvant therapys.

Participants must have a diagnosis of Diabetes Mellitus and Diabetic Foot; one or two chronic active ulcers at the time of assessment; and clinical levels of stress or anxiety or depression. Participants will be randomized by the four conditions - EG1, EG2, ACG and PCG - and assessed on the day of the first consultation or nursing treatment for chronic DFU (T0), two months later (T1), and six months later (T2; follow-up). Two weeks after T1, an interview will be conducted independently with patients that completed the relaxation, hypnosis, and placebo sessions, and with the informal caregivers who provided them the DFU care. The results of the present study will contribute for a better understanding of DFU progression, healing, prevention of re-ulceration and future amputations and, consequently, for the improvement of patients' quality of life.

DETAILED DESCRIPTION:
General Aim:

This RCT aims to assess the effectiveness of a muscle relaxation intervention with guided imagery (EG1) compared to hypnosis with guided imagery intervention (EG2) and a neutral guided imagery placebo (ACG) and a group that does not receive any psychological intervention (PCG), in DFU healing, physiological indicators of healing prognosis, and quality of life (QoL), in patients with diabetic foot and a chronic ulcer.

This study will also examine, qualitatively, the perspectives of patients and their respective family caregivers regarding the interventions (EG1 and EG2) and placebo sessions in order to check the treatments' effectiveness.

Specific aim:

1. To compare the impact of both experimental groups (EG1 and EG2) on psychological stress markers, in DFU healing, physiological indicators of healing prognosis, and QoL compared to the (PCG); between pre and post-intervention in the EG1 and EG2, controlling for clinical and sociodemographic variables, adherence to DFU care, and patients' literacy.

   Nested qualitative study specific aims:
2. To understand the perspectives of patients and family caregivers on the efficacy of EG1 and EG2 interventions versus ACG sessions to the DFU healing, comparing cases with a positive evolution (healing of the DFU) with cases with a negative evolution (DFU non-healing).

Sample size calculation:

Using Sakpal formula (2010), and according to the descriptive results of the pilot study (Ferreira et al., 2022), considering the difference in the mean (1.93) and standard deviation (6) of the treatment versus passive control groups, with a statistical power of 80% and a statistical significance level of 5%, a definitive RCT will require 152 participants. Considering a dropout rate for intervention sessions of 11%, a definitive RCT with four groups will require a sample of 169 participants, with 42 patients per group (Ferreira et al., 2022).

Procedure:

The doctor or nurse, in the medical appointment, identifies patients that meet the medical inclusion criteria. Patients are invited to participate in the study by the Researcher at the end of the medical appointment and are informed about the aims of the study and the voluntary nature of participation through an informed and informative consent. If patients agree to participate, they will sign the consent form. Nurses will then complete RESVECH 2.0 at the end of the appointment and doctors will complete the clinical questionnaire. Afterward, the Researcher will accompany the patient to a room provided by the Hospital in order to administer the battery of questionnaires in the interview format.

After answering the questionnaires, the researcher will score the PSS and HADS instruments to confirm the presence of significant clinical levels of stress, anxiety or depression, and if the patient is eligible, at the end of that week, the participant will be randomized into one of four possible groups.

In the next diabetic foot appointment, the respective participant will be informed about the group to which he or she has been allocated and whether will benefit, if appropriate, from four sessions of relaxation (EG1), hypnosis (EG2), or neutral guided imagery (ACG). If allocated to the PCG, the patient will not receive any psychological or placebo session. If the participant is available, the first session will take place on the same day. The following sessions will be scheduled according to the medical diabetic foot consultations. In each session, two assessments of blood pressure and heart rate will be performed, before starting the session and at the end of the session. At the end of the fourth session, the T1 assessment will be performed, with a new administration of the questionnaires. Six months after T0, the T2 (follow-up) evaluation will take place, with the last administration of the questionnaires. At T0, T1 and T2 a blood and DFU swab sample will be collected for the evaluation of the physiological variables. Plasma and peripheral blood mononuclear cells (PBMC)s will be separated from the blood samples and frozen at -80ºC for analysis by the biochemical team member. Blood lymphocyte populations will be analyzed by flow cytometry and the quantification of blood cell populations will be performed by an automated hematological cell counter on fresh blood samples. The medical and nurse team member, as well as the lab technicians will not be aware of which group participants belong to.

The interviews with patients who completed the four sessions of EG1, EG2, and ACG, as well as their informal caregivers, will be conducted separately, two weeks after T1, by a different researcher than the one involved in the sessions conduction, to reduce the bias of social desirability.

Data analysis:

All standard statistical analyses will be done using the Rstudio, R version 3.6.2 (R Core Team, 2019) and the SPSS statistics, v. 24.0 (IBM SPSS Statistics for Windows, IBM Corp, Armonk, New York). The baseline data of the treatments and control groups will be compared, using chi-squared test for binary variables and the t-test for continuous variables. The comparison between experimental groups (EG1 and EG2) and control groups (ACG and PCG) will be analyzed through Generalized Mixed Models.

A semi-structured interview guide consisting of open-ended questions will be administered to approximately 12 patients that benefited from interventions (EG1, EG2) and placebo (ACG) sessions), and 12 informal caregivers indicated by those patients. This script will remain unchanged throughout the interviews. The audio recording of the interviews will be done using a tablet, transcribed verbatim, and anonymized in order to safeguard participants and data confidentiality. The transcripts of the interviews will be analyzed in the same order as conducted, using the thematic content analysis technique, and the NVivo software (QSR International PtyLtd, 2018).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* Diabetes Mellitus diagnosis;
* Diagnosis of Diabetic Foot;
* Having one or two active chronic ulcers (> 6 weeks and < 14 weeks) at the time of baseline assessment;
* Being followed at the Multidisciplinary Consultation of the Diabetic Foot from the Centro Hospitalar Universitário do Porto (CHUP), at the Diabetic Foot Clinic from the Centro Hospitalar do Tâmega e Sousa (CHTS) and from the Multidisciplinary Consultation of the Diabetic Foot of the Hospital de Braga (HB);
* Presenting clinical levels of stress (scores > 13 for males and > 17 for females on the Perceived Stress Scale) or anxiety or depression (scores > 11 on Hospital Anxiety and Depression Scale);
* Providing written informed consent.

Exclusion Criteria:

* The active DFU at the time of the assessment being a relapse;
* Having more than two DFUs at the time of baseline assessment;
* Being on hemodialysis treatment;
* Presence of psychosis or dementia described in the patient's medical record;
* Having cancer disease;
* Having undergone a transplant;
* Receiving psychological counselling at the time of the assessment.

For the RCT qualitative nested study, twelve participants that completed at least 75% of the treatment or placebo sessions, and that report having a informal/ family caregiver will be invite the participate. Participants will be selected according to the following criteria:

* Two typical cases of successful and unsuccessful patients with neuropathic foot, defined by the presence of neuropathic pain (e.g., heat, tingling, electrical shock), presence of distal pulses by palpation, and loss of protective sensitivity;
* Two typical cases of successful and unsuccessful patients with neuroischemic foot, defined by the presence of peripheral artery disease, intense-variable pain, absence of distal pulses by palpation, and variable protective sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Impact of the DFU on patients' quality of life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The Diabetic Foot Ulcer Scale-Short Form (DFS-SF; Bann, Fehnel, & Gagnon, 2003; Research version by Pereira et al., 2022) will be used to assess patients´ DFU-related quality of life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better DFU-related quality of life.
Degree of DFU healing | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The degree of DFU healing will be assessed with the Portuguese version of "Resultados esperados de la valoración y evolución de la cicatrización de las heridas crónicas" Scale [Expected results of the evaluation and evolution of the healing of chronic wounds Scale - RESVECH 2.0] (Marques, 2015). The scores range from 0 to 35, where zero indicates complete healing.
Physical quality of life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The Short-Form Health Survey (SF-36; Ferreira, 1998; Ferreira, Ferreira, & Pereira, 2012) will be administered to assess patients' physical health-related quality of life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better physical quality of life.
Mental quality of life | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The Short-Form Health Survey (SF-36; Ferreira, 1998; Ferreira, Ferreira, & Pereira, 2012) will be administered to assess patients' mental health-related quality of life. Raw scores are transformed into a scale from 0 to 100. Higher results correspond to better mental quality of life.
Metabolic marker | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The quantification of HbA1c in the plasma will be performed using the competitive inhibition enzyme immunoassay Cloud Clone Corp
Inflammatory markers | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  IL-6, IL-8, and TNF-a levels will be evaluated in the plasma using a LEGENDplexTM Human Angiogenesis Panel 1 Mix and Match (9-plex). Blood lymphocyte populations will be assessed in the whole blood by flow cytometry and automated hematological cell counter.
Angiogenic markers | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Angiopoietin-2, EGF, FGF-basic, PECAM-1, PIGF, and VEGF levels will be assessed in the plasma using a LEGENDplexTM Human Angiogenesis Panel 1 Mix and Match (9-plex).
miRNA markers | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  miRNA-21 and miRNA-155 will be assessed with SYBR Green technology, using the RNU6B gene as control.
Immune cells | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Blood leukocyte and B and T-cell populations will be assessed in the whole blood by flow cytometry and automated hematological cell counter.

SECONDARY OUTCOMES:
Perceived Stress | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The overall stress perceived by the patient will be assessed through the Perceived Stress Scale (PSS; Trigo, Canudo, Branco, & Silva, 2010). Scores range between 0 and 40, with higher results indicating higher levels of perceived stress.
Emotional Distress | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The emotional distress will be assessed through the total score of the Hospital Anxiety and Depression Scale, comprising both anxiety and depression scales (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 42, with higher results indicating higher levels of distress.
Anxiety symptoms | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The anxious symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of anxiety symptoms.
Depression symptoms | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The depressive symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of depression symptoms.
Representations regarding the DFU | Changes from baseline (T0) to the end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Patient representations regarding the DFU will be evaluated through the Illness Perception Questionnaire - Brief (IPQ-B; Figueiras et al., 2010). The response scale ranges from 0 to 10. Higher scores indicate more threatening representations regarding DFU.

OTHER OUTCOMES:
Sociodemographic data | Baseline (T0)
  The following socio-demographic data will be collected: gender; age; living environment; marital status; professional status; monthly income; if there is an informal caregiver, what is the degree of kinship with the caregiver and the quality of the patient's relationship with the caregiver; as well as some questions regarding access to health care.
Clinical data | Baseline (T0), end of intervention/ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  The clinical data collected through a clinical questionnaire developed for this study will be: alcohol and tobacco consumption, presence and intensity of ulcer-related pain, and other symptomatic foot complaints; the type and duration of diabetes, HbA1c levels, duration of diabetic foot ulcer, type of foot and type of ulcer (PEDIS classification), location of the ulcer, recognised complications and comorbidities, type of treatment provided at the consultation, number of medical and nursing visits, date of DFU healing, and appearance of new ulcers. Psychophysiological parameters such as transcutaneous O2 pressure (TCPO2) where appropriate.
Health literacy | Baseline (T0)
  The level of health literacy will be assessed through the Medical Term Recognition Test (METER; Paiva et al., 2014).
Systolic pressure | Before and after each intervention session at week 2 (1st session), week 4 (2nd session), week 6 (3rd session), and week 8 (4th session). Also, after the baseline (T0), end of interv./ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Systolic pressure in millimeters of mercury (mmHg) will be assessed through a validated and certified blood pressure measuring device.
Diastolic pressure | Before and after each intervention session at week 2 (1st session), week 4 (2nd session), week 6 (3rd session), and week 8 (4th session). Also, after the baseline (T0), end of interv./ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Diastolic pressure in millimeters of mercury (mmHg) will be assessed through a validated and certified blood pressure measuring device.
Heart rate | Before and after each intervention session at week 2 (1st session), week 4 (2nd session), week 6 (3rd session), and week 8 (4th session). Also, after the baseline (T0), end of interv./ 2 months later at post-test (T1), and after 6 months follow-up (T2)
  Heart rate in beats per minute (bpm) will be assessed through a validated and certified blood pressure measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: M. Graça Pereira, PhD, Study Director — School of Psychology, University of Minho
Locations (3):
- Portugal (3):
  - Hospital de Braga, Braga
  - Clínica do Pé Diabético, Centro Hospitalar do Tâmega e Sousa, Penafiel
  - Centro Hospitalar Universitário do Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bann CM, Fehnel SE, Gagnon DD. Development and validation of the Diabetic Foot Ulcer Scale-short form (DFS-SF). Pharmacoeconomics. 2003;21(17):1277-90. doi: 10.2165/00019053-200321170-00004. PMID 14986739
- [Background] Bardin L. Análise de Conteúdo [Content Analysis]. 2016; São Paulo, Brasil: Almedina. Brasil.
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Direção-Geral de Saúde, DGS [General Health Direction, Portugal] Circular Normativa Nº:05/PNPCD: Pé Diabético, Programa Nacional de Prevenção e Controlo da Diabetes (PNPCD) [Normative Circular Nº: 05 / PNPCD: Diabetic Foot, National Diabetes Prevention and Control Program]; 2010. Retrieved from http://www.dgs.pt/?cr=15718
- [Background] Ferreira P. A medição do estado de saúde: Criação da versão portuguesa do MOS SF-36 [Measuring health status: Creation of the Portuguese version of MOS SF-36]. Coimbra: Centro de Estudos e Investigação em Saúde, Faculdade de Economia, Universidade de Coimbra; 1998. Ferreira PL, Ferreira LN, Pereira LN. Medidas sumário física e mental de estado de saúde para a população portuguesa [Physical and mental summary measures of health state for the Portuguese population]. Revista Portuguesa de Saúde Pública. 2012;30(2):163-171. doi:10.1016/j.rpsp.2012.12.007.
- [Background] Ferreira V, Martins J, Loureiro L, Loureiro T, Borges L, Silveira D, … Almeida R. Consulta multidisciplinar do pé diabético: Avaliação dos fatores de mau prognóstico [Multidisciplinary consultation of diabetic foot - factors related with bad prognosis]. Angiologia e Cirurgia Vascular. 2014;10:146-150. doi:10.1016/ j.ancv.2014.08.005
- [Background] Figueiras M, Marcelino DS, Claudino A, Cortes MA, Maroco J, Weinman J. Patients' illness schemata of hypertension: the role of beliefs for the choice of treatment. Psychol Health. 2010 Apr;25(4):507-17. doi: 10.1080/08870440802578961. PMID 20204931
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] International Working Group on the Diabetic Foot [IWGDF] International Consensus on the Diabetic Foot. International Diabetes Foundation; 2015. Retrieved from http://www.iwgdf.org/files/2015/website_prevention.pdf
- [Background] Marques JM. Adaptação cultural e validação para a população portuguesa de um instrumento de monitorização de feridas crónicas - escala RESVECH 2.0 [Cultural adaptation and validation for the Portuguese population of a chronic wound monitoring instrument - RESVECH 2.0 scale] (Master's Thesis). Instituto de Ciências da Saúde da Universidade Católica, Porto; 2015.
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Paiva D, Silva S, Severo M, Ferreira P, Santos O, Lunet N, Azevedo A. Cross-cultural adaptation and validation of the health literacy assessment tool METER in the Portuguese adult population. Patient Educ Couns. 2014 Nov;97(2):269-75. doi: 10.1016/j.pec.2014.07.024. Epub 2014 Jul 22. PMID 25107513
- [Background] Pandis N. Randomization. Part 3: allocation concealment and randomization implementation. Am J Orthod Dentofacial Orthop. 2012 Jan;141(1):126-8. doi: 10.1016/j.ajodo.2011.09.003. No abstract available. PMID 22196195
- [Background] Spiegel H. An eye-roll test for hypnotizability. Am J Clin Hypn. 1972 Jul;15(1):25-8. doi: 10.1080/00029157.1972.10402206. No abstract available. PMID 4679812
- [Background] Trigo M, Canudo N, Branco F, Silva D. Estudo das propriedades psicométricas da Perceived Stress Scale (PSS) na população Portuguesa [Psychometric proprieties of the Perceived Stress Scale (PSS) in Portuguese population]. Psychologica. 2010;53:353-378. doi:10.14195/1647-8606_53_17
- [Background] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Background] Ferreira G, Faria S, Carvalho A, Pereira MG. Relaxation intervention to improve diabetic foot ulcer healing: Results from a pilot randomized controlled study. Wound Repair Regen. 2023 Jul-Aug;31(4):528-541. doi: 10.1111/wrr.13085. Epub 2023 May 9. PMID 37078427